CLINICAL TRIAL: NCT03328052
Title: Randomized Trial Evaluating the Effectiveness of MYnd Analytics Directed Therapy in Depression
Brief Title: MYnd Analytics Directed Therapy in Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cota Inc. (Industry)
Collaborators: Hackensack Meridian Health (Other); Horizon Blue Cross Blue Shield of New Jersey (Other); MYnd Analytics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MYnd 001
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: All patients undergo EEG, but results are not released to physician or patient in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MYnd Analytics PEER Online directed therapy (Experimental): Patients in this arm will receive anti-depressants as recommended by the PEER Online algorithm as described below.
  Interventions: Device: MYnd Analytics PEER Online directed antidepressant therapy
- Conventional therapy (Sham Comparator): Patients in this arm will receive anti-depressants as chosen by the physician without guidance by the PEER Online algorithm.
  Interventions: Other: Conventional antidepressant therapy

INTERVENTIONS:
Device: MYnd Analytics PEER Online directed antidepressant therapy — PEER Online is similar to a standard QEEG in that it uses QEEG output variables, but differs from a standard QEEG in that it references the QEEG to a normative and then symptomatic database. By comparing a given patient's QEEG to a database of QEEGs of subjects who have tried and responded to a specific medication, PEER Online can provide useful information regarding the response of neuro-physiologically similar patients to a wide number of medications. PEER Online may thus have the advantage of providing physicians with useful information as to medication outcomes before a medication regime is started. It has also been used to help select the medication that best matches the QEEG brainwave pattern, regardless of "symptom clusters," currently used for diagnostic nomenclature. Patients will receive anti-depressant therapy guide by the results of the PEER Online algorithm.
  Arms: MYnd Analytics PEER Online directed therapy
Other: Conventional antidepressant therapy — Anti-depressant therapy chosen based on physician best judgement.
  Arms: Conventional therapy

SUMMARY:
The MYnd Analytics PEER Online strategy utilizes EEG diagnostics to direct patients with psychiatric illnesses to the best medication treatments. This trial will evaluate patients with a diagnosis of depression who will either receive (1) PEER Online directed therapy or (2) conventional treatment without EEG guidance and will compare 6 month clinical and economic outcomes between these groups.

DETAILED DESCRIPTION:
Mynd Analytics has developed the Psychiatric Electroencephalography Evaluation Registry (PEER) Online® clinical decision support database that uses a combination of software, analytics, and clinical outcomes to provide objective, adjunctive medication response information to physicians treating patients with non-psychotic behavioral disorders. PEER Online uses a statistical analysis of EEG outputs and other patient information to generate a report that indicates the statistical likelihood of the patient's responsiveness to classes of central nervous system (CNS) medications (i.e. antidepressants), groups (i.e. SSRI) and individual agents (i.e. fluoxetine). A discriminant analysis compares neurophysiologic abnormalities of the patient to patterns of abnormalities of known responders to CNS drugs in the company's outcomes database of symptomatic patients. This provides a probability estimate of the similarity of the patient's profile with the profile of groups of individuals constituting the normative and clinical (symptomatic) database, which provides the treating physician guidance to which treatments the patient will most likely respond to, and those treatments to which the patient is least likely to respond.

Procedurally, PEER Online utilizes standard 21-lead digital electroencephalographic equipment measuring the patient in a resting (but awake) state. The recording generally takes 30-60 minutes. Patients are classified based upon the 1,142 variables calculated in the recording (FDA-approved neurometric system) and categorized based on the outcome history in treating patients with similar neurophysiologic outputs. From these outputs and the correlation to the outcome database, reports may indicate single or multiple medications based on the nature of the physiologic abnormality discovered. The entire procedure is rapid, non-invasive, devoid of radiation or high strength magnetic fields, and results in a report, the PEER Outcome Report that is provided to clinicians in a format similar to antibiotic sensitivity testing.

Study Design (summary)

1. The patient population will consist of individuals with depression who in the opinion of their physician require medication management. A score of 10 or more on the PHQ-9 instrument will be required for enrollment. Non-psychotic co-morbid illnesses will be permitted. Patients must not currently be receiving psychotropic medications (including stimulants, benzodiazepines, or THC). Patients previously on these medications but off treatment for >30 days are permitted.
2. The physician will declare whether they wish to treat the depression or refer to a participating psychiatrist. Individual physicians (prior to enrolling any patients) will be assigned to either agree to utilize MYnd Analytic directed care or to be part of the control cohort. This will minimize any physician learning effect.
3. The patient will sign informed consent to participate.
4. All patients will undergo a study related EEG and MYnd Analytics will develop a PEER Online report. The report will be released to the treating physicians in the directed care group but will not be released to the control physicians.
5. All patients will complete a disease specific assessment tool (QIDS-SR16) at every office visit (at a minimum assessments at baseline, 3 months into treatment, and 6 months into treatment). Patients choosing to withdraw from the study or from treatment will also be offered the assessment at participation endpoint. COTA will score each patient based on the standardized tools as either improved, stable, or worsened. The primary endpoint for this study is QIDS-SR16 percent mean change from baseline, with response being defined as a reduction of >50% from baseline. Physicians may know the results of these tests and may alter therapy per their usual practice.
6. Medication management will be at the final discretion of the treating physician. Physicians assigned to the MYnd Analytics directed care cohort will be encouraged, but not required, to follow the PEER Online report. Any change in therapy will be documented by the physician with reason (lack of efficacy, toxicity, patient preference).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of depression who in the judgement of their physician require medication management may be eligible for enrollment. A score of 10 or more on the PHQ-9 instrument will be required for enrollment.
* Some practices utilize the PHQ-2 and PHQ-9 are part of routine screening for depression. If the tests are performed routinely, they do not need to be repeated for study eligibility, and may be performed prior to informed consent for this study. If, however, the PHQ-9 is not routinely performed, informed consent must be performed prior to administration. Patients with a score below 10 will be considered screen failures and will not be enrolled or offered the MYnd testing.
* Patients with non-psychotic comorbid conditions may be included.
* Patients must be either medication treatment naïve for behavioral illnesses or have no active medication treatments for at least 1 month prior to enrollment. Prohibited medications at the time of enrollment will include stimulants, benzodiazepines and THC. Prior therapy with these agents is permitted with a washout of >30 days.
* Patients must have private medical insurance coverage through Horizon Blue Cross Blue Shield. This is limited to insured commercial members, including HMO, and excluding, for the avoidance of doubt, members of self-insured customers or Medicare or Medicaid programs.

Exclusion Criteria:

* Diagnosis of a psychotic disorder.
* History of, or current, open head brain trauma. Candidates with any metal, shrapnel or other similar objects in the head that could affect the QEEG
* History of: craniotomy, cerebral metastases, cerebrovascular accident; current diagnosis of seizure disorder, schizophrenia, schizo-affective disorder, dementia, mental retardation, or major depression with psychotic features; or use of depot neuroleptics in last 12 months.
* Uncontrolled thyroid disorders.
* Known pregnancy and/or lactation, or intent to become pregnant during this study.
* Chronic or acute pain requiring prescription pain medication(s) (narcotic or synthetic narcotic)
* Participation in any other therapeutic drug study within 60 days preceding inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
50% Reduction From Baseline in Self-rated Severity of Depressive Symptoms as Measured by Quick Inventory of Depressive Symptomatology Self-Rated 16-item Scale (QIDS-SR-16) | 6 months
  QIDS-SR-16 is a 16-question self-report inventory that includes the 9 Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria symptom domains: sad mood, concentration, self-outlook, suicidal ideation, involvement, energy/fatigability, sleep disturbance (4 items: initial, middle, late insomnia, and hypersomnia), appetite/weight increased or decrease (4 items), and psychomotor agitation/retardation (2 items). The QIDS-SR-16 total scores range from 0 (least severe) to 27 (most severe). This study will examine the percentage of patients with improvement in depression as assessed by the QIDS-SR-16 at the 6 month treatment visit [repeated measures from all visits - for patients who received the intervention ie. MD followed PEER recommended therapy]. Response will be defined as a >50% reduction in QIDS-SR-16 score from baseline.

SECONDARY OUTCOMES:
Clinical improvement based on physician access to MyND Analytic PEER Online report. | 6 months
  Percentage of patients improving on the standardized assessments stratified by whether the physician had access to the MyND Analytic PEER Online report.
Persistence of PEER recommended therapy. | 3 months
  Percentage of patients remaining on PEER Online concordant therapy vs discordant therapy at the 3 month visit. Sub-analysis will include whether the patient was on the original therapy or whether changes were made due to lack of efficacy or toxicity. Switches in medications from a PEER recommended therapy to another recommended therapy based on a physician assessment of lack of efficacy will be counted as a failure, however a switch for toxicity will not be counted as failure.

OTHER OUTCOMES:
Total cost of care. | 6 months
  Total cost of care (all cause) for patients on PEER Online concordant therapy vs discordant therapy. Sub-analysis will focus on total cost of care based on whether the physician had access to the PEER report.
Exploring use of Cota Nodal Address (CNA) | 6 months
  CNA is a unique prognostic classification schema. All patients will undergo classification at time of diagnosis and exploratory analysis for patterns of responsiveness will be undertaken.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Solhkhah, MD, Principal Investigator — Hackensack Meridian Health
Locations (13):
- United States (13):
  - Hackensack Meridian Health Network, Brick, New Jersey
  - Hackensack Meridian Health Network, Hackensack, New Jersey
  - Hackensack Meridian Health Network, Holmdel, New Jersey
  - Hackensack Meridian Health Network, Jackson, New Jersey
  - Hackensack Meridian Health Network, Lodi, New Jersey
  - Hackensack Meridian Health Network, Neptune City, New Jersey
  - Hackensack Meridian Health Network, Oakhurst, New Jersey
  - Hackensack Meridian Health Network, Old Bridge, New Jersey
  - Hackensack Meridian Health Network, Paramus, New Jersey
  - Hackensack Meridian Health Network, Point Pleasant, New Jersey
  - Hackensack Meridian Health Network, Saddle Brook, New Jersey
  - Hackensack Meridian Health Network, Tinton Falls, New Jersey
  - Hackensack Meridian Health Network, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MYnd Analytics — http://www.mynd.com
- See also: COTA Healthcare — http://www.cotahealthcare.com